CLINICAL TRIAL: NCT03924986
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Compare the Efficacy and Safety of Tislelizumab (BGB-A317) Combined With Gemcitabine Plus Cisplatin Versus Placebo Combined With Gemcitabine Plus Cisplatin as First-Line Treatment for Recurrent or Metastatic Nasopharyngeal Cancer
Brief Title: Tislelizumab Combined With Chemotherapy Versus Chemotherapy Alone in Recurrent or Metastatic Nasopharyngeal Cancer (NPC)
Acronym: RATIONALE-309
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGB-A317-309; CTR20182534 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2019-03-21; First posted 2019-04-23 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Cancer
MeSH Terms: conditions — Recurrence; Nasopharyngeal Neoplasms | interventions — tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Tislelizumab + Gemcitabine + Cisplatin (Experimental): Participants received tislelizumab 200 mg intravenously (IV) once every 3 weeks (Q3W), gemcitabine 1 g/m^2 IV on days 1 and 8 of each 21-day cycle and cisplatin 80 mg/m^2 IV on day 1 of each cycle for 4 to 6 treatment cycles. Participants may have received treatment for longer at the Investigator's discretion until disease progression. Participants with confirmed disease progression may have continued to receive tislelizumab monotherapy.
  Interventions: Drug: Tislelizumab; Drug: Gemcitabine; Drug: Cisplatin
- Arm B: Placebo + Gemcitabine + Cisplatin (Placebo Comparator): Participants received placebo IV once every 3 weeks, gemcitabine 1 g/m^2 IV on days 1 and 8 of each 21-day cycle and cisplatin 80 mg/m^2 IV on day 1 of each cycle for 4 to 6 treatment cycles. Participants may have received treatment for longer at the Investigator's discretion until disease progression. Participants with confirmed disease progression may have crossed over to receive tislelizumab 200 mg IV Q3W monotherapy.
  Interventions: Drug: Placebo; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Tislelizumab — 200 mg intravenously (IV) once every 3 weeks (Q3W)
  Other Names: BGB-A317
  Arms: Arm A: Tislelizumab + Gemcitabine + Cisplatin
Drug: Placebo — Placebo to match tislelizumab (administered intravenously Q3W)
  Arms: Arm B: Placebo + Gemcitabine + Cisplatin
Drug: Gemcitabine — 1 gram per square meter of body surface area (g/m^2) on Day 1 and day 8 of each cycle, administered as an IV infusion within 30 minutes, for 4 to 6 cycles
Drug: Cisplatin — 80 milligrams per square meter of body surface area (mg/m^2) on Day 1 of each cycle, administered as an IV infusion for over 4 hours if possible or with proper infusion time based on local clinical guidelines or clinical practice and according to the treating physician's clinical judgment, for 4 to 6 cycles.

SUMMARY:
This study was designed to compare the efficacy and safety of tislelizumab (BGB-A317) combined with gemcitabine plus cisplatin versus placebo combined with gemcitabine plus cisplatin as first-line treatment for recurrent or metastatic nasopharyngeal cancer.

ELIGIBILITY:
Key Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
2. Aged between 18 to 75 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place)
3. Histologically or cytologically confirmed, recurrent or metastatic NPC
4. Participants must be able to provide fresh or archival tumor tissues (formalin-fixed paraffin-embedded [FFPE] blocks or approximately 10 [≥ 6] freshly cut unstained FFPE slides) with an associated pathological report. The archival tumor tissues must be collected within 2 years before screening. In the absence of sufficient archival tumor tissues, a fresh biopsy of a tumor lesion at baseline is mandatory
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Must have ≥ 1 measurable lesions as defined per RECIST v1.1
7. Must be treatment-naive for recurrent or metastatic NPC.

Key Exclusion Criteria:

1. Participants with locally recurrence suitable for curative surgery or radiotherapy
2. Received any approved systemic anticancer therapy, including hormonal therapy, within 28 days prior to initiation of study treatment. The following exception is allowed:

   * Palliative radiotherapy for bone metastases or soft tissue lesions should be completed > 7 days prior to baseline imaging.
3. Has received any immunotherapy (including but not limited to interferons, interleukin 2, tumor necrosis factor interleukin, and thymoxin) or any investigational therapies within 14 days or 5 half-lives (whichever is longer) of randomization
4. Received prior therapies targeting programmed cell death protein-1 (PD-1) or programmed cell death protein ligand-1 (PD-L1)
5. Active leptomeningeal disease or uncontrolled, untreated brain metastasis
6. Active autoimmune diseases or history of autoimmune diseases that may relapse
7. Any active malignancy ≤ 2 years before randomization except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- China (30):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The Peoples Hospital of Zhongshan City, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital Sun Yat Sen University, Zhuhai, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Taiwan (3):
  - Changhua Christian Hospital, Changhua
  - Veterans General Hospital Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
- Thailand (4):
  - Ramathibodi Hospital Mahidol University Hematology, Bangkok
  - Songklanagarind Hospital (Prince of Songkhla University), Hat Yai
  - Srinagarind Hospital (Khon Kaen University), Muang
  - Maharaj Nakorn Chiang Mai Hospital (Chiang Mai University), Muang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Zhang L, Liu T, Wang H, Shi S, Yang Y. A Phase 3 Trial in Progress Comparing Tislelizumab Plus Chemotherapy With Placebo Plus Chemotherapy in Chinese Patients With Recurrent or Metastatic Nasopharyngeal Cancer. Abstract published at: 22nd Annual Meeting of the Chinese Society of Clinical Oncology; September, 2019; Xiamen, China.
- [Derived] Yang Y, Pan J, Chen N, Guo Y, Huang X, Wu Y, Leaw S, Bai F, Wang Y, Zhao N, Tang B, Barnes G. Effects of tislelizumab on health-related quality of life in patients with recurrent or metastatic nasopharyngeal cancer. Head Neck. 2024 Sep;46(9):2301-2314. doi: 10.1002/hed.27785. Epub 2024 Apr 26. PMID 38671587
- [Derived] Yang Y, Pan J, Wang H, Zhao Y, Qu S, Chen N, Chen X, Sun Y, He X, Hu C, Lin L, Yu Q, Wang S, Wang G, Lei F, Wen J, Yang K, Lin Z, Guo Y, Chen S, Huang X, Wu Y, Liang L, Chen C, Bai F, Ma X, Zhang Y, Leaw S, Zhang L, Fang W. Tislelizumab plus chemotherapy as first-line treatment for recurrent or metastatic nasopharyngeal cancer: A multicenter phase 3 trial (RATIONALE-309). Cancer Cell. 2023 Jun 12;41(6):1061-1072.e4. doi: 10.1016/j.ccell.2023.04.014. Epub 2023 May 18. PMID 37207654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in multiple study centers in China, Thailand, and Taiwan. The first participant was consented on March 27th 2019, and the last participant completed on December 8th 2023.
Groups:
- Arm B: Placebo + Gemcitabine + Cisplatin: Participants received placebo IV once every 3 weeks, gemcitabine 1 g/m^2 IV on days 1 and 8 of each 21-day cycle and cisplatin 80 mg/m^2 IV on day 1 of each cycle for 4 to 6 treatment cycles. Participants may have received treatment for longer at the Investigator's discretion until disease progression. Participants with disease progression confirmed by the Independent Review Committee (IRC) may have crossed over to receive tislelizumab 200 mg IV Q3W monotherapy.
Period: Overall Study
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Started | 131 | 132
Treated | 131 | 132
Crossed Over to Tislelizumab | 0 | 70 (Includes one participant who crossed over to receive tislelizumab monotherapy but did not have IRC-confirmed disease progression.)
Completed | 0 | 0
Not Completed | 131 | 132
Not completed — Death | 57 | 66
Not completed — Study Concluded by Sponsor | 51 | 41
Not completed — Withdrawal by Subject | 15 | 20
Not completed — Lost to Follow-up | 7 | 5
Not completed — Miscellaneous | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) analysis set included all participants randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 131 | 132 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (10.62) | 49.5 (10.76) | 49.3 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 103 | 103 | 206
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 122 | 126 | 248
  Thailand | 5 | 1 | 6
  Taiwan | 4 | 5 | 9
Baseline Target Lesions Sum of Diameters Assessed by Investigator (mm) [Mean (Standard Deviation); unit: Millimeters (mm)] | 65.49 (49.004) | 57.56 (40.389) | 61.51 (44.978)

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival as Assessed by the Independent Review Committee (IRC)
Description: Defined as the time from randomization to the first objectively documented disease progression, or death from any cause, whichever occurred first, as assessed by the IRC per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Kaplan-Meier methodology was used to estimate the median PFS.
Time Frame: Through the study interim data analysis cutoff date of March 26th, 2021 (maximum time on study follow-up was 23 months)
Population: ITT analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 131 | 132
Months | 9.2 [7.6 to 10.1] | 7.4 [5.6 to 7.5]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Gemcitabine + Cisplatin vs Arm B: Placebo + Gemcitabine + Cisplatin; The null hypothesis to be tested is that progression-free survival (PFS) in Arm A is less than or equal to PFS in Arm B. This is compared against the alternative hypothesis, which posits that PFS in Arm A is greater than PFS in Arm B; Test type: Other; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.38 to 0.73] — Estimated using a Cox proportional hazards model with Efron's method for tied events, with Arm B as the reference group. The analysis was stratified by gender and liver metastases status

2. Secondary Outcome: Overall Response Rate (ORR) as Assessed by the IRC
Description: Defined as the percentage of participants who had complete response or partial response as assessed by the IRC per RECIST v1.1 in all randomized participants with measurable disease at Baseline.
Time Frame: Through the study interim data analysis cutoff date of March 26th, 2021 (maximum time on study follow-up was 23 months)
Population: ITT analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 131 | 132
percentage of participants | 69.5 [60.8 to 77.2] | 55.3 [46.4 to 64.0]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Gemcitabine + Cisplatin vs Arm B: Placebo + Gemcitabine + Cisplatin; Test type: Other; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.11 to 3.07]; Arm B was the reference group, and the odds ratio between arms was calculated using the Cochran-Mantel-Haenszel chi-square test, stratified by gender and liver metastases status

3. Secondary Outcome: Duration of Response (DOR) as Assessed by the IRC
Description: Defined as the time from the first occurrence of a documented objective response to the time of relapse, or death from any cause, whichever occurred first, as assessed by the IRC per RECIST v1.1 in all randomized participants with documented objective responses.
Time Frame: Through the study interim data analysis cutoff date of March 26th, 2021 (maximum time on study follow-up was 23 months)
Population: ITT analysis Set. Only participants with best overall response of complete response or partial response confirmed per RECIST v1.1 were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 91 | 73
months | 8.5 [6.5 to NA] — Not estimable due to insufficient number of participants with events | 6.1 [4.7 to 6.2]

4. Secondary Outcome: Overall Survival (OS) as Assessed by the IRC
Description: Defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: Through study completion data cut-off date of December 8th, 2023 or last available date showing participants alive (maximum time on study follow-up was 53 months)
Population: ITT analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 131 | 132
Months | 45.3 [33.4 to NA] — Not estimable due to insufficient number of participants with events | 31.8 [25.0 to NA] — Not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Gemcitabine + Cisplatin vs Arm B: Placebo + Gemcitabine + Cisplatin; Test type: Other; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.51 to 1.05] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: PFS as Assessed by the Investigator
Description: Defined as the time from randomization to the first objectively documented disease progression, or death from any cause, whichever occurred first, as assessed by the investigator per RECIST v1.1.
Time Frame: Through the interim analysis data cut-off date of March 26th, 2021 (up to approximately 23 months)
Population: ITT analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 131 | 132
months | 9.8 [7.8 to 11.9] | 7.6 [6.6 to 7.8]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab + Gemcitabine + Cisplatin vs Arm B: Placebo + Gemcitabine + Cisplatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.38 to 0.76] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Progression-free Survival After Next Line of Treatment (PFS2) as Assessed by the Investigator
Description: Defined as the time from randomization to second/subsequent disease progression after initiation of new anticancer therapy, or death from any cause, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Through the study completion data cut-off date of December 8th, 2023 (maximum time on study follow-up was 53 months)
Population: ITT analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 131 | 132
months | 45.3 [31.5 to NA] — Not estimable due to insufficient number of participants with events | 20.5 [13.9 to 27.2]

7. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status
Description: Change from baseline in EORTC QLQ-C30 Global Health Status/Quality of Life score. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of participants with cancer. It includes global health status and quality of life questions related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes.
Time Frame: Baseline to Cycle 6 (Each cycle is 21 days)
Population: The HRQoL analysis set includes all randomized participants who received any dose of study drug and completed at least one HRQoL assessment. Only participants with data at both baseline and the each postbaseline visit are included in the summary statistics for change from baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 108 | 104
score on a scale | 0.2 (25.18) | -0.1 (20.72)

8. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck-351 (EORTC QLQ-H&N35) Index Score
Description: The QLQ-H&N35 consists of thirty-five questions that are associated with eighteen symptom scales (pain, swallowing, senses, speech, social eating, social contact, sexuality, problem with teeth, problem opening mouth, dry mouth, problem with sense smell, cough, felt ill, pain med, nutritional supplements, feeding tube, weight loss and weight gain).. Raw scores are transformed into a 0 to 100 scale via linear transformation. The index score is calculated as an average of the 18 symptom scales. A negative change from baseline score indicates improvement in symptoms.
Time Frame: Baseline to Cycle 6 (Each cycle is 21 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 108 | 104
score on a scale | -0.3 (6.40) | -0.3 (7.17)

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory tests, vital signs, electrocardiograms (ECGs), and physical examinations (PEs ), graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. For Arm B, only adverse events reported prior to participants crossing over to receive tislelizumab monotherapy are included.
Time Frame: From first dose to 30 days after last dose or new anticancer therapy, or until Dec 8, 2023 data cut-off; max treatment duration: 231 weeks (Arm A), 202 weeks (Arm B).
Population: The Safety analysis set includes all randomized participants who received any dose of any component of study drug. Two participants randomized to Arm B who received 100 mg tislelizumab in error were analyzed as part of Arm A for the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin
Number analyzed (Participants) | 133 | 130
Participants
  TEAEs | 133 | 129
  SAEs | 47 | 46

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after the last dose or initiation of a new anticancer therapy, maximum duration of treatment was 231 weeks in Arm A and 202 weeks in Arm B.
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events include all randomized participants who received ≥ 1 dose of any study treatment. Two participants randomized to Arm B who received 100 mg tislelizumab in error were analyzed as part of Arm A for the Safety Analysis Set.
Groups:
- Post Crossover Tislelizumab: Participants in Arm B crossed over to receive tislelizumab 200 mg IV Q3W upon confirmed disease progression per RECIST v1.1 by the IRC, and with medical monitor approval.
Arm/Group | Arm A: Tislelizumab + Gemcitabine + Cisplatin | Arm B: Placebo + Gemcitabine + Cisplatin | Post Crossover Tislelizumab
All-Cause Mortality (participants affected / at risk) | 57/133 | 31/130 | 35/70
Serious Adverse Events (participants affected / at risk) | 47/133 | 46/130 | 15/70
Other Adverse Events (participants affected / at risk) | 133/133 | 129/130 | 60/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tislelizumab + Gemcitabine + Cisplatin (N=133) | Arm B: Placebo + Gemcitabine + Cisplatin (N=130) | Post Crossover Tislelizumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (4) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Accidental death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 1 (2)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 4 (5) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 6 (8) | 0 (0)
Platelet count decreased (Investigations) | 9 (12) | 14 (16) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 5 (6) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tislelizumab + Gemcitabine + Cisplatin (N=133) | Arm B: Placebo + Gemcitabine + Cisplatin (N=130) | Post Crossover Tislelizumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 114 (273) | 117 (235) | 19 (40)
Leukopenia (Blood and lymphatic system disorders) | 46 (281) | 44 (204) | 2 (6)
Myelosuppression (Blood and lymphatic system disorders) | 4 (5) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 46 (218) | 38 (159) | 1 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (51) | 16 (43) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 2 (2) | 5 (5) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 4 (5) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 11 (12) | 8 (8) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 5 (5) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 41 (70) | 20 (23) | 11 (15)
Abdominal discomfort (Gastrointestinal disorders) | 9 (19) | 8 (12) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 18 (25) | 15 (19) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 9 (14) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 9 (17) | 0 (0)
Constipation (Gastrointestinal disorders) | 46 (108) | 60 (130) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 21 (26) | 14 (28) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 17 (21) | 6 (9) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (7) | 3 (4) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 7 (9) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 10 (23) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 78 (206) | 94 (263) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 5 (10) | 7 (9) | 1 (1)
Toothache (Gastrointestinal disorders) | 9 (11) | 4 (4) | 6 (9)
Vomiting (Gastrointestinal disorders) | 55 (122) | 68 (175) | 4 (4)
Asthenia (General disorders) | 13 (17) | 11 (12) | 1 (1)
Chest discomfort (General disorders) | 9 (11) | 8 (12) | 1 (1)
Chest pain (General disorders) | 4 (4) | 2 (2) | 0 (0)
Fatigue (General disorders) | 17 (28) | 17 (26) | 1 (1)
Influenza like illness (General disorders) | 4 (6) | 4 (6) | 2 (3)
Malaise (General disorders) | 29 (70) | 31 (62) | 5 (5)
Non-cardiac chest pain (General disorders) | 4 (7) | 4 (5) | 2 (2)
Oedema peripheral (General disorders) | 5 (5) | 8 (15) | 0 (0)
Pyrexia (General disorders) | 34 (46) | 13 (20) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (2) | 4 (12) | 1 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (12) | 6 (10) | 0 (0)
COVID-19 (Infections and infestations) | 4 (7) | 1 (4) | 7 (13)
Nasopharyngitis (Infections and infestations) | 5 (6) | 4 (4) | 3 (4)
Otitis media (Infections and infestations) | 7 (7) | 2 (3) | 3 (3)
Periodontitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 22 (32) | 12 (15) | 6 (9)
Urinary tract infection (Infections and infestations) | 6 (7) | 4 (4) | 1 (2)
Alanine aminotransferase increased (Investigations) | 36 (59) | 26 (41) | 11 (11)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 7 (11) | 2 (2) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 38 (65) | 30 (47) | 11 (14)
Blood albumin decreased (Investigations) | 5 (5) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 8 (11) | 4 (8) | 3 (3)
Blood bilirubin increased (Investigations) | 8 (22) | 8 (10) | 1 (2)
Blood cholesterol increased (Investigations) | 4 (9) | 2 (2) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 4 (4) | 2 (2) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 11 (22) | 3 (4) | 6 (11)
Blood creatinine increased (Investigations) | 32 (60) | 22 (41) | 5 (8)
Blood lactate dehydrogenase increased (Investigations) | 13 (21) | 8 (9) | 3 (5)
Blood thyroid stimulating hormone increased (Investigations) | 8 (11) | 7 (8) | 3 (3)
Blood urea increased (Investigations) | 9 (18) | 8 (10) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 5 (7) | 2 (3) | 0 (0)
Fibrin D dimer increased (Investigations) | 4 (5) | 4 (4) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 9 (11) | 4 (8) | 3 (3)
Granulocyte count decreased (Investigations) | 4 (8) | 2 (5) | 0 (0)
Haemoglobin decreased (Investigations) | 5 (6) | 2 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 19 (52) | 23 (63) | 3 (13)
Monocyte count decreased (Investigations) | 7 (12) | 4 (4) | 0 (0)
Monocyte percentage decreased (Investigations) | 4 (6) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 80 (294) | 76 (306) | 6 (20)
Neutrophil count increased (Investigations) | 4 (4) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 68 (160) | 76 (202) | 1 (1)
Platelet count increased (Investigations) | 6 (13) | 5 (10) | 0 (0)
Red blood cell count decreased (Investigations) | 5 (8) | 3 (3) | 1 (2)
Thyroxine free decreased (Investigations) | 3 (3) | 2 (3) | 3 (3)
Weight decreased (Investigations) | 19 (20) | 14 (15) | 1 (2)
White blood cell count decreased (Investigations) | 81 (393) | 81 (454) | 8 (28)
Decreased appetite (Metabolism and nutrition disorders) | 64 (119) | 65 (132) | 4 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (13) | 4 (7) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (13) | 4 (4) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 (18) | 6 (12) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 24 (74) | 25 (53) | 7 (23)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 22 (39) | 29 (44) | 8 (17)
Hypocalcaemia (Metabolism and nutrition disorders) | 25 (40) | 17 (31) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 16 (28) | 22 (46) | 2 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (10) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 30 (47) | 29 (60) | 6 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 (44) | 16 (23) | 4 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 40 (75) | 36 (88) | 11 (13)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (18) | 8 (15) | 2 (11)
Hypoproteinaemia (Metabolism and nutrition disorders) | 12 (18) | 7 (10) | 3 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (32) | 17 (20) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (42) | 18 (22) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (11) | 5 (6) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 10 (12) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (22) | 10 (10) | 2 (3)
Dizziness (Nervous system disorders) | 22 (42) | 19 (35) | 2 (2)
Headache (Nervous system disorders) | 15 (22) | 22 (35) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 20 (37) | 20 (32) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 14 (17) | 17 (25) | 2 (2)
Haematuria (Renal and urinary disorders) | 4 (5) | 2 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 4 (6) | 1 (1)
Renal impairment (Renal and urinary disorders) | 5 (6) | 3 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (39) | 13 (16) | 11 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 12 (14) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 3 (3) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 17 (34) | 10 (23) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 2 (2) | 3 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 10 (13) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 10 (10) | 5 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 11 (11) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (74) | 18 (33) | 6 (9)
Rash (Skin and subcutaneous tissue disorders) | 34 (54) | 29 (34) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (8) | 4 (7) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 6 (7) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 4 (4) | 0 (0)
Phlebitis (Vascular disorders) | 4 (4) | 5 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT03924986/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT03924986/SAP_001.pdf